CLINICAL TRIAL: NCT02006186
Title: Pilot Study on Bicycle Trains to Improve Children's Physical Activity
Brief Title: Pilot and Feasibility Bicycle Train Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Jason Mendoza, Associate Professor of Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21HL113810 (NIH)
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Physical Activity
Keywords: Bicycling
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bicycle Train Intervention (Experimental): The Bicycle Train intervention consists of research staff members who bike to and from school with enrolled participants. All participants, regardless of group assignment, each receive a bicycle, safety equipment, and take a bicycle safety course.
  Interventions: Behavioral: Bicycle Train
- Control (No Intervention): The control arm does not receive any intervention. All participants, regardless of group assignment, each receive a bicycle, safety equipment, and take a bicycle safety course.

INTERVENTIONS:
Behavioral: Bicycle Train — The Bicycle Train intervention consists of research staff members who bike to and from school with enrolled participants
  Arms: Bicycle Train Intervention

SUMMARY:
US children's active commuting to school (ACS; walking or cycling to school), previously common (48% in 1969) is now uncommon (13% in 2009). This decline coincided with the obesity epidemic, which disproportionately affects low-income and ethnic minority children. Programs to increase children's moderate-to-vigorous physical activity (MVPA) and lower obesity and related chronic disease risk are necessary. The Bicycle Train is an innovative program in which children cycle to and from school led by adults. Bicycle Trains provide another option for ACS, especially for children who live too far to walk to school. No randomized controlled trials (RCT) have evaluated Bicycle Trains and children's ACS or MVPA. Increasing the percent of children who cycle to school is sub-objective PA-14 of US Healthy People 2020.

The Primary Goals are to (a) conduct a pilot cluster RCT of a Bicycle Train program among low-income, ethnic minority 4th and 5th grade children and (b) collect concurrent accelerometer and GPS data and validate algorithms to identify and measure physical activity intensity and duration for children's cycling compared to heart rate monitors.

Our Specific Aims will be to:

SA1) evaluate among 80 4th and 5th grade ethnic minority children the feasibility of a pilot cluster RCT of a Bicycle Train program for (a) recruiting participants for a planned full-scale cluster RCT (b) promoting their participation, and (c) identifying barriers/facilitators to their participation; and SA2) validate algorithms examining concurrent accelerometry and global positioning system (GPS) data to identify and measure children's physical activity intensity and duration while cycling compared to the criterion standards of heart rate monitoring and direct observation

Feasibility Criteria (FC): As recommended for pilot studies, in which the main goal is to test feasibility of a research protocol, a fully powered R01-funded cluster RCT will be determined to be feasible if:

FC 1) We successfully recruit 80 low-income 4th and 5th grade children for the pilot Bicycle Train cluster RCT FC 2) The intervention children participate in the Bicycle Train program on average twice/week or more FC 3) Algorithms analyzing concurrent GPS and accelerometer data have high agreement, i.e. >90% agreement, with heart rate data/direct observation in distinguishing children's cycling-related physical activity duration and intensity from other physical activities and riding in a motor vehicle

DETAILED DESCRIPTION:
Physical activity decreases the risk of cardiovascular disease, Type 2 Diabetes, and multiple cancers, and is important for obesity prevention. US children's active commuting to school (ACS; walking or cycling to school), previously common (48% in 1969) is now uncommon (13% in 2009). This decline coincided with the obesity epidemic, which disproportionately affects low-income and ethnic minority children. Programs to increase children's moderate-to-vigorous physical activity (MVPA) and lower obesity risk are necessary. The Bicycle Train is an innovative program in which children cycle to and from school led by adults. Bicycle Trains provide another option for ACS, especially for children who live too far to walk to school. No randomized controlled trials (RCT) have evaluated Bicycle Trains and children's ACS or MVPA. Increasing the percent of children who cycle to school is sub-objective PA-14 of US Healthy People 2020.

The Primary Goals are to (a) conduct a pilot cluster RCT of a Bicycle Train program among low-income, ethnic minority 4th and 5th grade children and (b) collect concurrent accelerometer and GPS data and validate algorithms to identify and measure physical activity intensity and duration for children's cycling compared to heart rate monitors. This pilot study will provide feasibility data and extend the validity of quantifying cycling-related MVPA for a future fully-powered R01-funded Bicycle Train cluster RCT.

Our Specific Aims will be to:

SA1) evaluate among 80 4th and 5th grade ethnic minority children the feasibility of a pilot cluster RCT of a Bicycle Train program for (a) recruiting participants for a planned full-scale cluster RCT (b) promoting their participation, and (c) identifying barriers/facilitators to their participation; and SA2) validate algorithms examining concurrent accelerometry and global positioning system (GPS) data to identify and measure children's physical activity intensity and duration while cycling compared to the criterion standards of heart rate monitoring and direct observation

Feasibility Criteria (FC): As recommended for pilot studies, in which the main goal is to test feasibility of a research protocol, a fully powered R01-funded cluster RCT will be determined to be feasible if:

FC 1) We successfully recruit 80 low-income 4th and 5th grade children for the pilot Bicycle Train cluster RCT FC 2) The intervention children participate in the Bicycle Train program on average twice/week or more FC 3) Algorithms analyzing concurrent GPS and accelerometer data have high agreement, i.e. >90% agreement, with heart rate data/direct observation in distinguishing children's cycling-related physical activity duration and intensity from other physical activities and riding in a motor vehicle

This R21 application will provide important planning and methods validation targeted towards ethnic-minority children, the population at highest risk for childhood obesity in the US.

ELIGIBILITY:
Inclusion Criteria:

* attends a study school and is in the 4th or 5th grade,
* physically capable of riding a bicycle to and from school
* lives within approximately 2-miles of a study school
* has room at home to safely store a bicycle.

Exclusion Criteria:

* not in the 4th or 5th grade at a study school
* incapable of riding a bicycle to and from school
* lives beyond approximately 2-miles of a study school
* does not have room at home to safely store a bicycle

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Post-Intervention Bicycling to School | During weeks 3-5 of the intervention
  Mode of transport to school

SECONDARY OUTCOMES:
Pre-Intervention Moderate-to-vigorous physical activity (MVPA) | Baseline
  MVPA measured objectively by a combination of accelerometry and GPS data.
Post-Intervention Moderate-to-vigorous physical activity (MVPA) | During weeks 3-5 of the intervention
  MVPA measured objectively by a combination of accelerometry and GPS data.
Pre-Intervention Bicycling to School | Baseline
  Mode of transport to school

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Mendoza, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Mendoza JA, Haaland W, Jacobs M, Abbey-Lambertz M, Miller J, Salls D, Todd W, Madding R, Ellis K, Kerr J. Bicycle Trains, Cycling, and Physical Activity: A Pilot Cluster RCT. Am J Prev Med. 2017 Oct;53(4):481-489. doi: 10.1016/j.amepre.2017.05.001. Epub 2017 Jun 28. PMID 28668251